CLINICAL TRIAL: NCT03141073
Title: A 24-week Multi-center, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of HMS5552 add-on to Metformin With Additional 28-week Open-label Treatment to Evaluate the Safety in T2DM Subjects
Brief Title: Long-term Efficacy and Safety of HMS5552 add-on to Metformin in T2DM Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMM0302
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GKA; T2DM; HMS5552; Add-on therapy; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin; glucokinase activator compound 50

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMS5552 (Experimental): 75mg BID
  Interventions: Drug: HMS5552
- Placebo (Placebo Comparator): BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMS5552 — BID oral administration
  Other Names: Glucokinase Activator (GKA)
  Arms: HMS5552
Drug: Placebo — BID oral administration
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety and population PK of HMS5552 add-on to Metformin in adult type 2 diabetic subjects. There will be 2 groups in the first 24 weeks, one group will receive HMS5552 plus Metformin, while the other group will receive placebo plus Metformin; after 24 weeks, all subjects will receive HMS5552 plus Metformin for 28 weeks.

DETAILED DESCRIPTION:
This study is a phase III study in subjects with T2DM. As designed, the study will start with a 4-week, single-blind, placebo run-in period based on diet and exercise interventions for screening eligible subjects, meanwhile, subjects are treated with Metformin (Glucophage) at 1500mg/day as basic therapy throughout the treatment period. 3 weeks after run-in, eligibility is confirmed with required laboratory tests at -5±2 days prior to randomization. The eligible subjects are randomly assigned to HMS5552 75mg BID group or placebo BID group with ratio 1:1 to receive a 24-week double-blind treatment. Then all subjects receive 28-week open-label treatment of HMS5552 75mg BID add-on to Metformin. After 52-week treatment, all investigational drugs should be discontinued, followed by 1 week for safety evaluation. The dosage of Metformin (Glucophage) should be maintained at 1500 mg/day from run-in period to treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18~75 years old;
2. T2DM and treated with Metformin ≥ 1500mg/day constantly for at least 12 consecutive weeks;
3. 7.5% ≤ HbA1c ≤ 10.0% at screening;
4. 18.5 kg/m2 < BMI < 35.0 kg/m2 at screening;

Exclusion Criteria:

1. Any anti-diabetic therapy other than Metformin within 12 weeks before screening;
2. Received insulin therapy more than 30 days within 1 year before screening;
3. Fasting C-peptide <0.81 ng/ml (0.27 nmol/L) at screening;
4. Medical history of severe hypoglycemia or frequent hypoglycemia, diabetic ketoacidosis, diabetes lactic acidosis or hyperosmotic nonketotic diabetic coma, severe cardio-cerebrovascular, unstable or rapidly progressive kidney disease, active liver diseases, diagnosed mental disease etc.
5. T1DM;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 24 weeks
  The change of HbA1c from baseline by comparing HMS5552 75 mg BID in combination with Metformin with Placebo BID in combination with Metformin in T2DM subjects after 24-week double-blind treatment

SECONDARY OUTCOMES:
The change of 2-hour postprandial plasma glucose (2h-PPG) from baseline | 24 weeks
  The change of 2-hour postprandial plasma glucose (2h-PPG) from baseline by comparing HMS5552 75 mg BID in combination with Metformin with Placebo BID in combination with Metformin in T2DM subjects after 24-week double-blind treatment
The change of fasting plasma glucose (FPG) from baseline | 24 weeks
  The change of fasting plasma glucose (FPG) from baseline by comparing HMS5552 75 mg BID in combination with Metformin with Placebo BID in combination with Metformin in T2DM subjects after 24-week double-blind treatment
The proportion of subjects with HbA1c < 7.0% | 24 weeks
  HbA1c response rate by comparing HMS5552 75 mg BID in combination with Metformin with Placebo BID in combination with Metformin in T2DM subjects after 24-week double-blind treatment
The change of HbA1c from baseline at each visit over time, except at Week 24 | 24 weeks
  The change of HbA1c from baseline by comparing HMS5552 75 mg BID in combination with Metformin with Placebo BID in combination with Metformin in T2DM subjects at each visit over time, except at Week 24
Incidence of Treatment-Emergent Adverse Events over time | 52 weeks
  including incidence of adverse events, incidence of hypoglycemic events, physical examination, vital signs, 12-lead ECG, clinical laboratory examinations (routine blood test, blood biochemistry and routine urine test).

CONTACTS AND LOCATIONS:
Overall Officials: Wenying Yang, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Hua Medicine Limited, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang W, Zhu D, Gan S, Dong X, Su J, Li W, Jiang H, Zhao W, Yao M, Song W, Lu Y, Zhang X, Li H, Wang G, Qiu W, Yuan G, Ma J, Li W, Li Z, Wang X, Zeng J, Yang Z, Liu J, Liang Y, Lu S, Zhang H, Liu H, Liu P, Fan K, Jiang X, Li Y, Su Q, Ning T, Tan H, An Z, Jiang Z, Liu L, Zhou Z, Zhang Q, Li X, Shan Z, Xue Y, Mao H, Shi L, Ye S, Zhang X, Sun J, Li P, Yang T, Li F, Lin J, Zhang Z, Zhao Y, Li R, Guo X, Yao Q, Lu W, Qu S, Li H, Tan L, Wang W, Yao Y, Chen D, Li Y, Gao J, Hu W, Fei X, Wu T, Dong S, Jin W, Li C, Zhao D, Feng B, Zhao Y, Zhang Y, Li X, Chen L. Dorzagliatin add-on therapy to metformin in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled phase 3 trial. Nat Med. 2022 May;28(5):974-981. doi: 10.1038/s41591-022-01803-5. Epub 2022 May 12. PMID 35551292